CLINICAL TRIAL: NCT02366000
Title: A Randomized Controlled Trial of a Brief Intervention by Parents to Prevent Their Children From Experimenting With Health Risk Behavior: a Pilot Study
Brief Title: An Intervention Study: Shaping a Healthier Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hong Kong Sheng Kung Hui Tung Chung Integrated Services (Unknown)
Responsible Party: Principal Investigator, Dr. Yim Wah Mak, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AP-J86
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Parent-Child Relationship
Keywords: Parent-child communication; Health risk behaviors; Randomized controlled trial
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Parental Training Intervention (Experimental): Participants will have to attend two 3-hour Brief Parental Training Intervention Programme, with three weeks apart. There will also be two telephone follow-up sessions to reinforce learnt strategies and skills for home practice between workshops.
  Interventions: Other: Brief Parental Training Intervention
- Wait-list Group (Other): Participants will receive the same Brief Parental Training Intervention Programme as the intervention group. However, they will wait until the questionnaires have been completed by the intervention group for the second time (i.e. immediately after intervention) before they receive their programme.
  Interventions: Other: Brief Parental Training Intervention

INTERVENTIONS:
Other: Brief Parental Training Intervention — The workshop was designed to assist parents to communicate with their children about issues in the prevention of health risk behaviours- alcohol, tobacco and other drug use (ATOD), by equipping them with the appropriate interaction skills and encouraging them to build relationships with their children.

SUMMARY:
The aim of this study is to identify parent-children communication in relation to health risk behaviors (smoking, drinking and illegal drug taking) in adolescents, and to enhance better parental skills in preventing these behaviors in children.

DETAILED DESCRIPTION:
Previous research found that parent-children communication is the best predictor of health risk behaviors among adolescents. However, longitudinal studies of parent-adolescent communication on the subject of health risk behavior such as alcohol, tobacco and other drug use (ATOD) remain relatively scarce, and none of this kind of work has been done among Chinese sample. Such information is urgently needed given the increasing trend of drug use among adolescents in Hong Kong, and the severe burden of morbidity and mortality related to ATOD.

The study aims to examine parent-children communication in relation to health risk behaviors and to explore the potential efficacy of a brief intervention which is designed to assist parents of primary school children to communicate with their children about issues in the prevention of health risk behaviors. The efficacy of the intervention will be compared with a waiting-list control group using a randomized controlled trial. There will then be two telephone follow-ups to reinforce learnt strategies and skills for home practice in between the two workshops. There will also be assessments post-intervention and at 1 year follow-up. Evaluation focus groups will also be conducted after the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child in primary five or six
* Cantonese-speaking
* Consent to their participation in the program and the inclusion of their children in the assessments

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Readiness of parents to communicate with their children about preventing health risk behaviour | At 1 year
  Measured by Parent Questionnaire (PQ) - the sections on their (a) intention to take action, (b) self-efficacy in taking action, (c) plan of the action, (d) action to change (modified from Sniehotta, Scholz et al. 2002).

SECONDARY OUTCOMES:
Quality of parent-child communication | At 1 year
  Measured by Parent Questionnaire (PQ)- the section on parent-adolescent communication (Caprara, Pastorelli, Regalia, Scabini & Bandura, 2005) as well as the Chidren Questionnaire (CQ)- the section on parent-adolescent communication (Caprara et al, 2005)
Parents' attitudes towards positive parenting | At 1 year
  Measured by Parent Questionnaire (PQ)- the section on parenting patterns (Rohner, 1986; Chen, Rubin & Li, 1997)
Quality of parent-child relationships | At 1 year
  Measured by Parent Questionnaire (PQ)- the section on parent-child relationships (Schumm, Paff-Bergen et al., 1986) as well as the section on Children Questionnaire (CQ)- the section on parent-child relationships Schumm et al., 1986)
Children's health risk behaviour | At 1 year
  Measured by Children Questionnaire (CQ)- the sections on health risk behaviour - smoking (Mak et al, 2005; Abdullah et al, 2006); alcohol use (Ewing, 1984); and illicit drug use (Kolbe, Kann & Collins, 1999; Lee & Tsang, 2004)

CONTACTS AND LOCATIONS:
Overall Officials: YW Mak, PHD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University

REFERENCES:
- [Background] Caprara GV, Pastorelli C, Regalia C, Scabini & Bandura A. (2005). Impact of adolescents' Filial self-efficacy on quality of family functioning and satisfaction. Journal of Research on Adolescence. 15(1). 71-97.
- [Background] Rohner, R. P. (1984). Handbook for the study of parental acceptance and rejection (Rev. Ed.). Storrs: Center for the Study of Parental Acceptance and Rejection, University of Connecticut
- [Background] Schumm, W. R., Paff-Bergen, L. A., Hatch, R. C., Obiorah, F. C., Copeland, J. M., Meens, L. D., et al. (1986). Concurrent and Discriminant Validity of the Kansas Marital Satisfaction Scale. Journal of Marriage and the Family, 48,381-387.
- [Background] Sniehotta, F.F., Scholz, U., Lippke, S. & Zielmann, J. (2002). Scale for assessment of implementation planning and coping planning. http://userpage.fu-berlin.de/~falko/scales/heartdocu.html
- [Background] Abdullah AS, Mak YW, Loke AY, Lam TH. Smoking cessation intervention in parents of young children: a randomised controlled trial. Addiction. 2005 Nov;100(11):1731-40. doi: 10.1111/j.1360-0443.2005.01231.x. PMID 16277633
- [Background] Mak YW, Loke AY, Lam TH, Abdullah AS. Validity of self-reports and reliability of spousal proxy reports on the smoking behavior of Chinese parents with young children. Addict Behav. 2005 May;30(4):841-5. doi: 10.1016/j.addbeh.2004.08.008. PMID 15833586
- [Background] Ewing JA. Detecting alcoholism. The CAGE questionnaire. JAMA. 1984 Oct 12;252(14):1905-7. doi: 10.1001/jama.252.14.1905. PMID 6471323
- [Background] Kolbe LJ, Kann L, Collins JL. Overview of the Youth Risk Behavior Surveillance System. Public Health Rep. 1993;108 Suppl 1(Suppl 1):2-10. No abstract available. PMID 8210269
- [Background] Lee A, Tsang CK. Youth risk behaviour in a Chinese population: a territory-wide youth risk behavioural surveillance in Hong Kong. Public Health. 2004 Mar;118(2):88-95. doi: 10.1016/S0033-3506(03)00174-4. PMID 15037037